CLINICAL TRIAL: NCT00429117
Title: Interest in Spirituality and Oncology: Is It An International Phenomenon?
Status: Withdrawn | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0724
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Stress
Keywords: Spirituality; Work Related Stress; Religious Beliefs; Survey
MeSH Terms: conditions — Occupational Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey: Physician members of the International Gynecologic Oncologists Society or the Society of Gynecologic Oncologists.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Internet survey lasting 30 to 40 minutes.
  Other Names: questionnaire

SUMMARY:
Primary Objective:

-To assess correlations between spiritual and religious beliefs and physician burnout using the Work Related Stress Inventory.

Secondary Objectives:

* To assess relationships between a physician's spiritual/religious beliefs and age, race, sex, marital status, and nationality.
* To explore differences in survey responses among oncologists from different countries: Duke University Religion Index (DUREL), Hoge (Intrinsic religiosity scale), Templer's Death Anxiety Scale, Locus of Control Scale, Work Related Strain Inventory, and non-validated case scenarios.
* To correlate survey responses to management of specific patient case situations.

DETAILED DESCRIPTION:
Few studies have explored the spiritual/religious beliefs of physicians and almost none have been done outside of the United States until the last two years. Therefore, this is the first study of its kind to evaluate this subject internationally.

In the next few weeks individuals will be receiving an on line survey from Survey Monkey.

The purpose of the survey is to explore the spiritual/religious beliefs of oncologists from a world side perspective, to identify areas in which spiritual/religious beliefs may affect medical decision making, and to explore any correlation that may exist between spiritual/religious beliefs of oncologists and physician burn out.

The surveys will take about 30 to 40 minutes to complete. Survey results will be encrypted even in transmission and sent to a secure server for anonymity. Even if one chooses not to fill out the surveys investigators ask that each person complete the demographic questionnaire.

Without input, investigators will lose the opportunity to further an understanding of how spirituality and religious beliefs impact patient care and physician well being.

Investigators welcome any feed back.

ELIGIBILITY:
Inclusion Criteria:

* Physician members of the International Gynecologic Oncologists Society or the Society of Gynecologic Oncologists

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physician members of the International Gynecologic Oncologists Society or the Society of Gynecologic Oncologists.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Survey response to assess correlations between spiritual and religious beliefs and physician burnout. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org